CLINICAL TRIAL: NCT01397526
Title: Colloid Osmotic Pressure During Heart Surgery in Children
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Indrebo, Cand.med, Oslo University Hospital
Other Study IDs: 063.09 (REK); 21443(NSD) (Other: Norwegian Social Science Data Sevices)
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Heart Defects, Congenital
Keywords: Congenital heart disease; Cardiopulmonary bypass; Capillary leak; Colloid osmotic pressure; Children
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Interstitial fluid Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Clinical oedema is seen after open heart surgery with the use of cardiopulmonary bypass and hypothermia in children. The oedema formation is due to increased fluid transport from blood to tissue. This transcapillary fluid transport is dependent on differences in interstitial and plasma colloid osmotic pressure. The purpose of this investigation is to evaluate changes in interstitial colloid osmotic pressure before, under and after the use of cardiopulmonary bypass in children. The study hypothesis is that oedema developed during cardiopulmonary bypass and hypothermia is caused by increased micro vascular protein leakage and reduced colloid osmotic pressure gradient through the capillary membrane.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of a congenital heart defect
* scheduled for open heart surgery with the use of cardiopulmonary bypass
* under 13 year of age
* informed consent obtained from the parents

Exclusion Criteria:

* renal failure
* liver failure

Ages: 1 Day to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children scheduled for open heart surgery with the use of Cardiopulmonary Bypass at Oslo University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2011-07; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Interstitial colloid osmotic pressure | Before, during and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Norgard, Prof. PhD, Study Chair — Oslo University Hospital; Ansgar Berg, Prof. PhD, Study Director — Haukeland University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway